CLINICAL TRIAL: NCT03432338
Title: Distribution of Non-Motor Symptoms in Idiopathic Parkinson's Disease and Secondary Parkinsonism A Controlled, Descriptive Cross-sectional Study Using Parkinson's Well-Being Map™
Brief Title: Distribution of Non-Motor Symptoms in Idiopathic Parkinson's Disease and Secondary Parkinsonism
Status: Completed | Type: Observational
Sponsor: Örjan Skogar (Other Government)
Responsible Party: Sponsor-Investigator, Örjan Skogar, MD,PhD, Region Jönköping County
Organization: Region Jönköping County (Other Government)
Other Study IDs: Dnr 2016/118-31
Record Dates: First submitted 2017-09-01; First posted 2018-02-14 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- idiopathic parkinson: Classical Parkinson´s disease, idiopathic
  Interventions: Other: inquiries
- secondary parkinsonism: parkinsonism due to other reasons than idiopathic
  Interventions: Other: inquiries
- controls: persona matched by age and gender, non parkinsonism
  Interventions: Other: inquiries

INTERVENTIONS:
Other: inquiries — Inquires reported to clinician.

SUMMARY:
BACKGROUND:

Non-Motor Symptoms (NMS) are frequent in patients with Idiopathic Parkinson's Disease (IPD). Clinical expressions, postulated pathophysiological mechanisms and responsiveness to antiparkinson medication represent differences between IPD and secondary Parkinsonism (SP).

OBJECTIVES:

To evaluate NMS expressions in IPD, SP and a control group.

METHODS:

Diagnosis of SP was supported by comorbidity, radiological findings, type of onset, onset rate and progression, exposures for neuroleptics, and responsiveness to pharmacological antiparkinson therapy.

The participants were consecutively recruited at two outdoor patient clinics. The Well-Being Map™ for evaluation. These were completed by the participants at one point before visit. The controls consisted of non-Parkinsonian individuals, matched by age and gender.

DETAILED DESCRIPTION:
Over the past decades knowledge of the natural history and progression of Parkinson´s disease (PD) has increased. Age at onset, time to troublesome complications are well described. Parallell to this, the society has been more and more aware of differences between gender in the expressions of diseases. Differences in self reported experiences are of great interest as this is tightly interconnected with Health Related Quality of Life, (HRQoL).

The incidence of PD rapidly increase over the age of 60 years (y) , with only 4% of the cases being under the age of 50 y. The rate for men 19.0 per 100,000, was 91% higher than that for women (9.9 per 100,000 )The age- and gender-adjusted rate per 100,000 was highest among Hispanics (16.6,non-Hispanic Whites ,Asians (11.3, and Blacks (10.2). These data suggest that the incidence of Parkinson's disease varies by race/ethnicity.

( ref. Van den Eeden 2003)

Nonmotor Symptoms in Parkinson's Disease:

Of the nine domains in the validated NMSS (Chaudhuri, Martinez- Martin, Brown, et al., 2007), sexual dysfunction and mood changes have been commonly observed to have associations with specific gender. While sexual dysfunction has been commonly reported with a significantly higher proportion among men (Kova ́cs, Makkos, Aschermann, et al., 2016; Martinez-Martin, Falup Pecurariu, Odin, et al., 2012; Picillo, Amboni, Erro, et al., 2013; Solla, Cannas, Ibba, et al., 2012; Szewczyk- Krolikowski, Tomlinson, Nithi, et al., 2014), mood symptoms, which encompass loss of interest in surroundings, lack of motivation, feeling ner- vous, flat mood, and difficulty in experiencing pleasure, have been frequently reported among women in a higher proportion compared to men with PD (Guo, Song, Chen, et al., 2013; Martinez-Martin et al., 2012; Nicoletti, Vasta, Mostile, et al., 2017; Solla et al., 2012; Song, Gu, An, & Chan, 2014).

It is well known that in the general population ( not specific parkinsonism ) in industrialized societies men die earlier than women but that women have poorer health than men. Differences discussed are differences in biological risks and acquired risks . But studies have revealed that the variations in health experiences depend on the particular symptom or condition in question and also according to the phase of the life cycle.

Already In an article by S.Macintyre et al from 1996 two large British surveys were examined and revealed a larger complexity than earlier studies had shown in the description of health surveys and differences between gender. These often described the consistency of reporting more illness , poorer self-evaluation of health and higher rates of psychosocial malaise in women than in men.

In this study more complex patterns of sex differences were shown for different symptoms reported. 'Worrying', 'nerves', 'always tired', 'headaches', 'constipation' and 'fainting or dizziness' showed the most consistent female excess. Sickness, nausea or stomach trouble were only dominating among 18 year old females and 'trouble with eyes' among 56-60 year olds in another large survey. In contrast, two symptoms, 'palpitations' and 'trouble with ears' show a male excess among middle aged. Female excess was only consistently found across the life span for the more psychological manifestations of distress, and was far less apparent for a number of physical symptoms and conditions.

Problems relating to reproduction will naturally show a female excess in the childbearing years, hormonal differences are apparent before and after the menopause.

Probably an oversimplification have been the fact in older sociological and epidemiological literature and over-generelization has become the norm.

There is a widely accepted belief that women use health services, particularly mental health services, more than men. Haavio-Manila has, however, reported that while women had higher psychiatric admission rates than men in Norway, in Finland and Sweden men had higher rates (Haavio-Manila E. Inequalities in health and gender. Soc. Sci. Med. 22, 141, 1986.) Why are more recent data more complex to understand than older studies in the field of gender differences? One possibility is that female/male differences in health have changed over time (in the same way that male/female differences in life expectancy may have changed over time (Macintyre S. Gender differences in longevity and health in Eastern and Western Europe. In Locating Health: Sociological and Historial Explanations (Edited by Platt S., Thomas H., Scott S. and Williams G.), pp. 57-74. Avebury, Aldershot, 1993.

If we are to make progress towards understanding to whether social, psychological or biological produce or maintain gender differences in health, it is important to pay attention to the social and historical context of the observations, and to take a more differentiated agespecific and condition-specific view of 'health' when examining differences between the sexes.

(Wingard D. L., Cohn B. A., Kaplan G. A., Cirillo P. M. and Cohen R. D. Sex differentials in morbidity and mortality risks examined by age and cause in the same cohort. Am. J. Epidemiol. 130, 601, 1989. )

National Quality Registers

A National Quality Registry contains individualised data concerning patient problems, medical interventions, and outcomes after treatment; within all healthcare production. It is annually monitored and approved for financial support by an Executive Committee.

Swedish Neuro Registries is a quality register with the aim of ensuring that neurological care is equitable and of high quality and to ensure treatment guidelines are being followed.

Swedish Neuro Registries are represented in all counties and all hospitals where neurological care is provided. It will be the base for national neurological research.

The registry started as an MS registry in 1996. In 2012, it became Swedish Neuro Registries with 8 diagnosis: Multiple Sclerosis, Parkinson's Disease, Myasthenia Gravis , Narcolepsy, Epilepsy, Motor Neuron Disease, Inflammatory Polyneuropathy and Severe Neurovascular Headache. REFERENS:( http://kvalitetsregister.se/englishpages/findaregistry/registerarkivenglish/nationalqualityregistryforneurologicalcareneuroregpreviouslyswedishmsregistry.2283.html Today abou 5800 patients are registered within the PD registry, of which about 4600 with a diagnose of PD or related disorders such as parkinsonism, atypical PD etcetera.

ELIGIBILITY:
Inclusion Criteria:

" Clinical diagnosis of Idiopathic Parkinson´s Disease " Clinical diagnosos of secondary parkinsonism " Healthy controls " Age >65 years " >1 year duration of disease after diagnose

Exclusion Criteria:

" Participation in other studies " Severe disease of psychiatric origin " Severe cognitive impairment

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Participants diagnosed with IPD or SP were recruited from routine care visits at outpatient departments at two medium-sized county hospitals in southern Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of selfreported motor and non-motor symptoms with The Parkinson´s Well-being map | 12 months
  A graded check list presented in The Parkinson´s Well-BeingMap is used in the registration of self reported frequencies and self experienced strength of Motor and Non- Motor Symptoms in two different forms of parkinsonism and in a group of healthy controls.The experienced magnitude of suffering is visualized in a spider diagram reflecting the strength of each item on an ordinal scale from 0 to four.
  Primary outcome measure is to compare reported frequencies between groups.

SECONDARY OUTCOMES:
Prevalence of combinations of reported motor and non-motor symptoms using | 12 months
  Secondary outcome measures are to study commonly reported combinations of non-motor symptoms within the groups, with respect to gender and duration of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Boel Andersson Gäre, PhD, Study Director — Region Jönköping County

IPD SHARING:
Plan to Share IPD: No